CLINICAL TRIAL: NCT06005415
Title: Glycemic Response to an Innovative Cookie to Promote Human Health
Acronym: GRINCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kristin Verbeke, Professor, KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: S67376
Record Dates: First submitted 2023-08-01; First posted 2023-08-22 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Postprandial Glycemic Responses
Keywords: postprandial glycemic responses; gastric emptying rate; oral processing behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test cookie (Active Comparator): Wire-cut cookie portion (85 g) containing wheat flour, coarse wheat semolina, sucrose, vegetable shortening, water, sodium chloride, sodium bicarbonate and sodium octanoate.
  Interventions: Dietary Supplement: Wire-cut cookie
- Control cookie (Active Comparator): Wire-cut cookie portion (85 g) containing wheat flour, wheat bran, sucrose, vegetable shortening, water, sodium chloride, sodium bicarbonate and sodium octanoate.
  Interventions: Dietary Supplement: Wire-cut cookie

INTERVENTIONS:
Dietary Supplement: Wire-cut cookie — Investigation of the impact of wheat particle size on the postprandial glycemic response, gastric emptying and oral processing behavior after consumption of wire-cut cookies.

SUMMARY:
The aim of this study is to investigate whether using a coarse wheat fraction in wire-cut cookie making induces a lower glycemic response in healthy subjects compared to wheat flour.

DETAILED DESCRIPTION:
This study has a double-blind, randomized, cross-over design. During each of the two study visits, healthy participants will consume a standard portion of cookies. One cookie formulation will present a large amount of coarse wheat fraction, while the other formulation will include only wheat flour and will serve as a control. Blood glucose measurements will be taken postprandially at regular time points. Gastric emptying rate and oral processing behavior will be also object of study.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) range 18.5 - 25.0 kg/m2 at screening visit
* Fasting whole blood glucose values < 6.3 mmol/L
* Regular diet with 3 meals a day (at least 5 times a week)
* Absence of health conditions that would prevent fulfillment of study requirements as judged by the Investigators on the basis of medical history
* Willingness to maintain habitual diet, physical activity pattern, and body weight throughout the trial
* Willingness to abstain from alcohol consumption and to avoid vigorous physical activity for 24 h prior to study visits
* Adequate level of understanding spoken and written English
* Willingness to report lifestyle factors such as level of physical activity and perceived psychological stress
* Willingness to provide informed consent to participate in the study

Exclusion Criteria:

* Failure to meet any one of the inclusion criteria
* Recent participation in any clinical trial (< 90 days)
* Pregnant or lactating or wishing to become pregnant in the period of the study
* Known history of AIDS, hepatitis, diabetes mellitus (Type I and II), cardiovascular disease, any pathology (or recent surgical event) of the gastrointestinal system or any current metabolic or endocrine disease
* Alcohol consumption of > 14 standard drinks for women and > 21 standard drinks for men per week
* Currently smoking (have smoked in the last 28 days) or willingness to smoke during the study period
* Celiac disease or gluten intolerance
* Use of medications known to influence carbohydrate metabolism, including, but not limited to adrenergic blockers, diuretics, thiazolidinediones, metformin and systemic corticosteroids the last 4 weeks before the screening visit
* Use of antibiotics during the last three months
* Reported slimming or medically prescribed diet
* Unwillingness or inability to comply with the experimental procedures and to follow the safety guidelines

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
Glucose response | 10, 5 minute before and 10, 20, 30, 45, 60, 75, 90, 120, 150 and 180 minutes after consumption of test meal, both test day 1 and 2
  Incremental area under the curve of blood glucose concentration (mM) after wheat-based wire-cut cookie consumption, measured through blood samples collected via finger-prick before eating (i.e. 10 and 5 minutes before ingestion) and at respective time points after consumption of test meal (i.e. 10, 20, 30, 45, 60, 75, 90, 120, 150 and 180 minutes).

SECONDARY OUTCOMES:
Peak rise of blood glucose | 10, 5 minute before and 10, 20, 30, 45, 60, 75, 90, 120, 150 and 180 minutes after consumption of test meal, both test day 1 and 2
  Difference between the highest postprandial blood glucose concentration and the baseline (expressed in mM), measured through blood samples collected via finger-prick before eating (i.e. 10 and 5 minutes before ingestion) and at respective time points after consumption of test meal (i.e. 10, 20, 30, 45, 60, 75, 90, 120, 150 and 180 minutes).
Gastric emptying rate | 0, 10, 20, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180 minutes after consumption of test meal, on test day 1
  Measured through 13C-octanoic acid breath samples collected before eating (i.e. 0 minute) and at respective time points after consumption of test meal (i.e. 10, 20, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180 minutes).
Gastric emptying rate | 0, 10, 20, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180 minutes after consumption of test meal, on test day 2
  Measured through 13C-octanoic acid breath samples collected before eating (i.e. 0 minute) and at respective time points after consumption of test meal (i.e. 10, 20, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180 minutes).
Oral processing behavior (exposure time) | During test meal consumption, up to 10 minutes, on test day 1
  Participants will be video-recorded to analyze oral processing behavior of the test meal. Number of bites, chews, swallows and time in mouth (s) will be annotated to derive total oral exposure time (s).
Oral processing behavior (exposure time) | During test meal consumption, up to 10 minutes, on test day 2
  Participants will be video-recorded to analyze oral processing behavior of the test meal. Number of bites, chews, swallows and time in mouth (s) will be annotated to derive total oral exposure time (s).
Oral processing behavior (average bite size) | During test meal consumption, up to 10 minutes, on test day 1
  Participants will be video-recorded to analyze oral processing behavior of the test meal. Number of bites, chews, swallows and time in mouth (s) will be annotated to derive total average bite size (g per bite).
Oral processing behavior (average bite size) | During test meal consumption, up to 10 minutes, on test day 2
  Participants will be video-recorded to analyze oral processing behavior of the test meal. Number of bites, chews, swallows and time in mouth (s) will be annotated to derive total average bite size (g per bite).
Oral processing behavior (average chews per bite) | During test meal consumption, up to 10 minutes, on test day 1
  Participants will be video-recorded to analyze oral processing behavior of the test meal. Number of bites, chews, swallows and time in mouth (s) will be annotated to derive total average chews per bite.
Oral processing behavior (average chews per bite) | During test meal consumption, up to 10 minutes, on test day 2
  Participants will be video-recorded to analyze oral processing behavior of the test meal. Number of bites, chews, swallows and time in mouth (s) will be annotated to derive total average chews per bite.
Oral processing behavior (eating rate) | During test meal consumption, up to 10 minutes, on test day 1
  Participants will be video-recorded to analyze oral processing behavior of the test meal. Number of bites, chews, swallows and time in mouth (s) will be annotated to derive total eating rate (g per minute).
Oral processing behavior (eating rate) | During test meal consumption, up to 10 minutes, on test day 2
  Participants will be video-recorded to analyze oral processing behavior of the test meal. Number of bites, chews, swallows and time in mouth (s) will be annotated to derive total eating rate (g per minute).
Oral processing behavior (energy intake rate) | During test meal consumption, up to 10 minutes, on test day 1
  Participants will be video-recorded to analyze oral processing behavior of the test meal. Number of bites, chews, swallows and time in mouth (s) will be annotated to derive total energy intake rate (kcal per minute).
Oral processing behavior (energy intake rate) | During test meal consumption, up to 10 minutes, on test day 2
  Participants will be video-recorded to analyze oral processing behavior of the test meal. Number of bites, chews, swallows and time in mouth (s) will be annotated to derive total energy intake rate (kcal per minute).

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Verbeke, Prof., Principal Investigator — KU Leuven
Locations (1):
- KU Leuven/UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No